CLINICAL TRIAL: NCT06307470
Title: Impact of a Nurse-led Mind-body Intervention on Sexual Health for Young Women
Brief Title: Nurse-led Mind-body Intervention on Sexual Health for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Intimate Pathways Center for Sexual Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 276879
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Women's Health: Neoplasm of Breast; Menopause, Premature; Body Image; Sexual Dysfunction; Cancer, Breast
Keywords: breast cancer; young women; cancer survivorship; sexual functioning; body image; premature menopause
MeSH Terms: conditions — Menopause, Premature; Sexual Dysfunction, Physiological; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMBRACE Group (Experimental): Immediately following consent, participants randomized to the EMBRACE Group will begin with the EMBRACE intervention. Participants will meet with a registered nurse certified in sexuality and sex education for 8 sessions every two weeks depending on scheduling. Each of the 8 sessions will last between 60 - 90 minutes. By session 2, participants will receive vaginal rehydration (Hyalo-Gyn suppositories), vaginal dilation (CalExotics Dr. Berman Dilator), and vaginal lubrication (Good Clean Love BioNude). These products will be mailed to participants at no cost to the participants.
  Participants will complete baseline measures, immediately following the intervention, and six weeks after the last session. Participants will be compensated for their time with a total up to $150.
  Interventions: Behavioral: EMBRACE (Empowerment through Mind and Body Reclamation After Cancer Experience)
- Delayed EMBRACE Group (Active Comparator): After consenting, participants randomized to the Delayed EMBRACE Group will begin with the EMBRACE intervention 16 weeks after enrollment. Participants will meet with a registered nurse certified in sexuality and sex education for 8 sessions every two weeks depending on scheduling. Each of the 8 sessions will last between 60 - 90 minutes. By session 2, participants will receive vaginal rehydration (Hyalo-Gyn suppositories), vaginal dilation (CalExotics Dr. Berman Dilator), and vaginal lubrication (Good Clean Love BioNude). These products will be mailed to participants at no cost to the participants.
  Participants will complete baseline measures, immediately following the intervention, and six weeks after the last session. Participants will be compensated for their time with a total up to $150.
  Interventions: Behavioral: EMBRACE (Empowerment through Mind and Body Reclamation After Cancer Experience)

INTERVENTIONS:
Behavioral: EMBRACE (Empowerment through Mind and Body Reclamation After Cancer Experience) — The intervention will be led by a registered nurse who holds certifications in sexuality counseling and sex education. The therapeutic, online environment will serve as a confidential, private space without judgement to encourage discussion to model safe sexuality communication for breast cancer survivors. The curriculum will include: i) psychoeducation: sexual body, mind-body connection, and sexual relationships; ii) physical-body education: physical response, safety, and navigating physical changes in survivorship; iii) solution-focused tools: tailored vaginal rehydration, lubrication, education; and iv) communication: internal, partnered, and patient-provider communication skills.
  The solution-focused tools will include vaginal rehydration and dilation products with vaginal lubrication. Tools will be distributed via mail by Session 2.

SUMMARY:
The goal of this clinical trial is to test the efficacy of a nurse-led psychoeducational sexual health intervention for young women breast cancer survivors. The main questions it aims to answer are:

1. What is the feasibility of this intervention in an online, private setting?
2. What is the effect of this intervention on reducing menopausal symptoms, improving sexual functioning, and enhancing body image?

Participants will participate in a nurse-led psychoeducational intervention for 8 sessions lasting approximately an hour each over the course of 16 weeks. Each participant will complete survey items at the beginning, end, and six-weeks after the last session. Participants will be compensated up to $150 in gift cards as a thank-you for their time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with breast cancer (stages I - III) between ages 18 - 50
* Completed active treatment (chemotherapy and/or radiation) within the last five years
* Can read/speak English
* Access to talk in quiet, safe environment for privacy
* On hormonal therapies (aromatase inhibitors, tamoxifen)
* Currently partnered (i.e., in a relationship)

Exclusion Criteria:

* Currently undergoing active treatment (chemotherapy and/or radiation)
* More than five years have passed since completing active treatment (chemotherapy and/or radiation)
* History of advanced breast cancer (stage IV) or a breast cancer recurrence
* Women without access to the internet
* Cannot read/speak in English

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on gender at birth.
Enrollment: 43 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Vulvovaginal Symptoms Questionnaire (VSQ) | Week 1, Week 16, Week 22
  A 21-item survey designed to measure vaginal symptoms, emotions, life impact due to vulvovaginal symptoms, and sexual impact of vulvovaginal symptoms. The scores range from 0 - 20 with the higher score meaning greater impact from vulvovaginal symptoms.
Body Image Scale | Week 1, Week 16, Week 22
  A 10-item survey designed to measure body image changes after cancer treatment. Scores range from 0 - 30 with the higher scores representing more body image disturbances related to cancer treatment.
Female Sexual Functioning Index | Week 1, Week 16, Week 22
  A 19-item survey measuring female sexual functioning. Scores range from 2 - 36 with the higher score representing greater sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Pearman D Parker, PhD, MPH, RN, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juraskova I, Jarvis S, Mok K, Peate M, Meiser B, Cheah BC, Mireskandari S, Friedlander M. The acceptability, feasibility, and efficacy (phase I/II study) of the OVERcome (Olive Oil, Vaginal Exercise, and MoisturizeR) intervention to improve dyspareunia and alleviate sexual problems in women with breast cancer. J Sex Med. 2013 Oct;10(10):2549-58. doi: 10.1111/jsm.12156. Epub 2013 May 1. PMID 23635341
- [Background] Wettergren L, Eriksson LE, Bergstrom C, Hedman C, Ahlgren J, Smedby KE, Hellman K, Henriksson R, Lampic C. Prevalence and risk factors for sexual dysfunction in young women following a cancer diagnosis - a population-based study. Acta Oncol. 2022 Oct;61(10):1165-1172. doi: 10.1080/0284186X.2022.2112283. Epub 2022 Sep 29. PMID 36176069
- [Background] Marsh S, Borges VF, Coons HL, Afghahi A. Sexual health after a breast cancer diagnosis in young women: clinical implications for patients and providers. Breast Cancer Res Treat. 2020 Dec;184(3):655-663. doi: 10.1007/s10549-020-05880-3. Epub 2020 Sep 23. PMID 32968951
- [Background] Rash JK, Seaborne LA, Peterson M, Kushner DM, Sobecki JN. Patient reported improvement in sexual health outcomes following care in a sexual health clinic for women with cancer. Support Care Cancer. 2023 Feb 16;31(3):171. doi: 10.1007/s00520-023-07635-4. PMID 36795172
- [Background] Esplen MJ, Wong J, Warner E, Toner B. Restoring Body Image After Cancer (ReBIC): Results of a Randomized Controlled Trial. J Clin Oncol. 2018 Mar 10;36(8):749-756. doi: 10.1200/JCO.2017.74.8244. Epub 2018 Jan 22. PMID 29356610
- [Background] Mifsud A, Pehlivan MJ, Fam P, O'Grady M, van Steensel A, Elder E, Gilchrist J, Sherman KA. Feasibility and pilot study of a brief self-compassion intervention addressing body image distress in breast cancer survivors. Health Psychol Behav Med. 2021 May 21;9(1):498-526. doi: 10.1080/21642850.2021.1929236. PMID 34104572
- [Background] Jun EY, Kim S, Chang SB, Oh K, Kang HS, Kang SS. The effect of a sexual life reframing program on marital intimacy, body image, and sexual function among breast cancer survivors. Cancer Nurs. 2011 Mar-Apr;34(2):142-9. doi: 10.1097/NCC.0b013e3181f1ab7a. PMID 20885305
- [Background] Panjari M, Bell RJ, Davis SR. Sexual function after breast cancer. J Sex Med. 2011 Jan;8(1):294-302. doi: 10.1111/j.1743-6109.2010.02034.x. Epub 2010 Sep 23. PMID 21199377
- [Background] Rosenberg SM, Vaz-Luis I, Gong J, Rajagopal PS, Ruddy KJ, Tamimi RM, Schapira L, Come S, Borges V, de Moor JS, Partridge AH. Employment trends in young women following a breast cancer diagnosis. Breast Cancer Res Treat. 2019 Aug;177(1):207-214. doi: 10.1007/s10549-019-05293-x. Epub 2019 May 30. PMID 31147983
- [Background] Ruddy KJ, Greaney ML, Sprunck-Harrild K, Meyer ME, Emmons KM, Partridge AH. A qualitative exploration of supports and unmet needs of diverse young women with breast cancer. J Community Support Oncol. 2015 Sep;13(9):323-9. doi: 10.12788/jcso.0169. PMID 26859752
- [Background] Vegunta S, Kuhle CL, Vencill JA, Lucas PH, Mussallem DM. Sexual Health after a Breast Cancer Diagnosis: Addressing a Forgotten Aspect of Survivorship. J Clin Med. 2022 Nov 14;11(22):6723. doi: 10.3390/jcm11226723. PMID 36431200
- [Background] Gorman JR, Drizin JH, Smith E, Flores-Sanchez Y, Harvey SM. Patient-Centered Communication to Address Young Adult Breast Cancer Survivors' Reproductive and Sexual Health Concerns. Health Commun. 2021 Nov;36(13):1743-1758. doi: 10.1080/10410236.2020.1794550. Epub 2020 Jul 23. PMID 32703034